CLINICAL TRIAL: NCT03106870
Title: Adding Metformin to Insulin in Controlling Pregestational and Gestational Diabetes Mellitus and Improving Neonatal Outcome Regarding Birth Weight
Brief Title: Adding Metformin to Insulin in Controlling Pregestational and Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Abdelrahman, Lecturer of Obstetrics and Gynaecology Faculty of Medicine, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Metformin
Record Dates: First submitted 2017-03-28; First posted 2017-04-11 (Actual); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
MeSH Terms: interventions — insulin, pork; isophane insulin, pork drug combination 30:70; Biphasic Insulins; Metformin

STUDY DESIGN:
Intervention Model Description: Group I: pregnant women who received oral metformin in addition to insulin therapy.
  Group II: pregnant women who received insulin therapy only.
Who Masked: Participant
Masking Description: Sixty-two opaque envelopes were numbered serially and in each envelope the corresponding letter which detect allocated group were put according to randomization then all envelops were closed and put in one box .When the first patient arrives , the first envelope were opened and the patient were allocated according to the letter inside .
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral metformin and insulin (Active Comparator): Intervention 'Insulin Mixtard' and Intervention 'metformin' had included
  Interventions: Drug: Insulin Mixtard; Drug: Metformin
- insulin therapy only (Active Comparator): Intervention 'Insulin Mixtard' had included
  Interventions: Drug: Insulin Mixtard

INTERVENTIONS:
Drug: Insulin Mixtard — Insulin dose:
  * 0.7 IU/Kg (at the second trimester of pregnancy).
  * 0.8 IU/Kg (at the third trimester of pregnancy). Insulin dose was raised at a rate of 1 IU for every 10 mg/dl higher than the target blood glucose concentration.
  Other Names: insulin mixtures
Drug: Metformin — Oral metformin at a dose of 1500 mg divided into three doses, were taken with meals, in addition to insulin.
  If the target blood glucose concentrations were not attained, the dose of metformin was raised to 2000 mg per day.
  Other Names: Metformin Hydrocloride
  Arms: oral metformin and insulin

SUMMARY:
The purpose of the study to prove benefits of adding metformin to insulin for controlling presentational and gestational diabetes mellitus and improving neonatal outcome.

DETAILED DESCRIPTION:
The current study was conducted at Ain Shams university maternity hospital during the period between June 2016 to December 2016.

All patients were subjected to:

1. History taking:
2. General and Abdominal Examination:

   With particular emphasis on :
   * Body mass index
   * Blood pressure.
   * Fundal height .
   * Estimated fetal weight .
3. Insulin and metformin doses :

   Insulin dose:

   0.7 IU/Kg (at the second trimester of pregnancy). 0.8 IU/Kg (at the third trimester of pregnancy). Insulin dose was raised at a rate of 1 IU for every 10 mg/dl higher than the target blood glucose concentration.

   Metformin dose :

   Oral metformin at a dose of 1500 mg divided into three doses, were taken with meals, in addition to insulin.

   If the target blood glucose concentrations were not attained, the dose of metformin was raised to 2000 mg per day.
4. Investigations:

Fasting and two hours postprandial blood glucose levels were measured in two groups of pregnant women:

1. Group I: pregnant women who received oral metformin in addition to insulin therapy.
2. Group II: pregnant women who received insulin therapy only.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 - 35 years.
2. Gestational age: 20- 36 weeks gestation.
3. Singleton pregnancy.
4. Women with pregestational or gestational diabetes mellitus

Exclusion Criteria:

1. Pregnant women with secondary diabetes (e.g. those on chronic steroid therapy).
2. Hypertensive patients.
3. Women with impaired liver or renal function
4. Non-compliant patients.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The current study was conducted at Ain Shams university maternity hospital during the period between June 2016 to December 2016.
  Sixty two pregnant women were recruited from Ain Shams university maternity hospital who fulfilled the inclusion criteria. They were counseled and after consenting were included into the study.
Groups:
- Oral Metformin and Insulin: Intervention 'Insulin Mixtard' and Intervention 'metformin' had included
  Insulin Mixtard: Insulin dose:
  * 0.7 IU/Kg (at the second trimester of pregnancy).
  * 0.8 IU/Kg (at the third trimester of pregnancy). Insulin dose was raised at a rate of 1 IU for every 10 mg/dl higher than the target blood glucose concentration.
  Metformin: Oral metformin at a dose of 1500 mg divided into three doses, were taken with meals, in addition to insulin.
  If the target blood glucose concentrations were not attained, the dose of metformin was raised to 2000 mg per day.
- Insulin Therapy Only: Intervention 'Insulin Mixtard' had included
  Insulin Mixtard: Insulin dose:
  * 0.7 IU/Kg (at the second trimester of pregnancy).
  * 0.8 IU/Kg (at the third trimester of pregnancy). Insulin dose was raised at a rate of 1 IU for every 10 mg/dl higher than the target blood glucose concentration.
Period: Overall Study
Arm/Group | Oral Metformin and Insulin | Insulin Therapy Only
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Metformin and Insulin | Insulin Therapy Only | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 31 | 62
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (3.9) | 29.7 (3.5) | 29.3 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Glycemic Control Over Period From 20 Weeks to 36 Weeks Gestation
Description: Fasting and two-hours postprandial blood glucose every 48 hours, till reaching the target blood glucose concentrations:
  60 - 95 mg/dl and < 120 mg/dl (for fasting and two-hour postprandial status, respectively) If patient reached blood glucose concentrations, she considered as controlled Diabetes Mellitus If patient did not reach blood glucose concentrations, she considered as uncontrolled Diabetes Mellitus
Time Frame: from 20 weeks to 36 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Metformin and Insulin | Insulin Therapy Only
Number analyzed (Participants) | 31 | 31
Participants | 24 | 27

2. Secondary Outcome: Number of Participants With a Macrosomic Baby
Description: Fetal macrosomia has been defined birth weight greater than 4500 gm
Time Frame: 24 hours after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Metformin and Insulin | Insulin Therapy Only
Number analyzed (Participants) | 31 | 31
Participants | 5 | 12

3. Secondary Outcome: Number of Participants With Neonates Who Were Hypoglycemic
Description: Neonatal hypoglycemia defined as a plasma glucose level of less than 30 mg/dL in the first 24 hours after delivery
Time Frame: 24 hours after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Metformin and Insulin | Insulin Therapy Only
Number analyzed (Participants) | 31 | 31
Participants | 5 | 6

ADVERSE EVENTS:
Time Frame: 7 months from June 2016 to December 2016
Description: Adverse Events of oral metformin and insulin were assessed.
Arm/Group | Oral Metformin and Insulin | Insulin Therapy Only
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No